CLINICAL TRIAL: NCT00201136
Title: Hypertension Improvement Project (HIP)
Brief Title: Interventions to Improve Hypertension Control and Reduce Cardiovascular Disease Risk
Acronym: HIP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Pro00013310; R01HL075373 (NIH)
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2015-10-14 (Estimated); Status verified 2012-02

CONDITIONS: Hypertension
Keywords: Behavioral intervention; Lifestyle modification; Guidelines
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- MD-C/PT-C (No Intervention): Physician and patient control group.
- MD-I/PT-C (Experimental): MD CQI-type intervention; Patient control
  Interventions: Behavioral: MD CQI-type intervention
- MD-C/Pt-I (Experimental): MD control; patient behavioral intervention
  Interventions: Behavioral: Lifestyle interventions to lower blood pressure for patients
- MD-I/Pt-I (Experimental): MD CQI-type intervention; Patient behavioral intervention
  Interventions: Behavioral: Lifestyle interventions to lower blood pressure for patients; Behavioral: MD CQI-type intervention

INTERVENTIONS:
Behavioral: Lifestyle interventions to lower blood pressure for patients — Weight loss, DASH dietary pattern, increased physical activity, reduced salt intake, moderation of alchohol intake.
  Arms: MD-C/Pt-I; MD-I/Pt-I
Behavioral: MD CQI-type intervention — CQI-type intervention for MD adherence to JNC guidelines for BP management
  Arms: MD-I/PT-C; MD-I/Pt-I

SUMMARY:
This study will test the separate and combined effects of a continuous quality improvement (CQI) intervention for physicians (MDs) and a behavioral intervention for patients on blood pressure control.

DETAILED DESCRIPTION:
BACKGROUND:

Hypertension affects 25% of adults in the United States and remains a leading cause of heart disease, stroke, and kidney failure. Despite numerous effective treatments, only 25% of people with hypertension are at goal blood pressure (BP). The chronic care model suggests that BP control can be achieved by improving patient self-care and the systems through which care is delivered. Patient self-care efforts should be directed at counteracting the effects of obesity, physical inactivity, poor dietary pattern, and non-adherence to prescribed medications on BP. In addition, efforts should be directed at the use of quality improvement systems that can counteract the well-documented non-adherence of primary care MDs to established clinical practice guidelines. In addition to improving BP control, these approaches can also reduce costs associated with hypertension and its consequences. However, given the resources that would be required to implement such approaches, it is critical that their effectiveness be rigorously established. This controlled study will test the separate and combined effects of a behavioral intervention for patients and a CQI intervention for MDs on BP control. The patient intervention will employ proven behavioral methods for promoting a healthy lifestyle and adherence to medication regimens. The MD intervention will use a CQI approach to provide training, motivation, and feedback on performance in a non-threatening way to promote continuous self-improvement and adherence to clinical practice guidelines.

DESIGN NARRATIVE:

The Hypertension Improvement Project (HIP) is a randomized, controlled study that will test the separate and combined effects of a CQI intervention for MDs and a behavioral intervention for patients on BP control. MDs will be selected from practices in the Duke Primary Care Research Consortium that serve low-income and minority populations. Practices will be randomly assigned to the MD intervention or to the MD control condition. Within these practices, all MDs will receive the same intervention and their patients will be individually randomized to the patient intervention or to the patient usual care condition. The MD intervention consists of the following three main elements: 1) on-line training modules; 2) an evaluation and treatment algorithm for use in the clinic; and 3) a CQI procedure involving assessment of clinical performance measures and feedback to MDs on their adherence to guidelines. The performance data will be collected for 18 months and feedback will be provided to MDs every 3 months. Patients from these practices (approximately 50% women, at least 40% African American, and 90% low-income) will be randomly assigned to patient intervention or usual care. The patient intervention consists of a 6-month behavioral intervention aimed at lifestyle changes to lower BP and promote adherence to prescribed BP medications. BP and other follow-up measurements will be performed at the end of the intervention and a year later (at 6 and 18 months post-randomization). The primary outcome will be the proportion of patients in each treatment group that have adequate BP control at 6 months. BP control is defined by the Joint National Committee 6 (JNC-6) goals (systolic BP less than 140 mm Hg and diastolic BP less than 90 mm Hg for most patients; lower goals for patients with cardiovascular or renal disease, or diabetes). Other outcomes of this study will include BP control at 18 months, MD adherence to national guidelines, and patient adherence to lifestyle recommendations and medication regimens. A cost analysis will also be done. The study will enroll 500 patients in 10 practices (approximately 20 MDs), and will have 80% power to detect an effect size of 0.3 for the primary outcome. The HIP study will test practical interventions for improving hypertension control that can be broadly implemented and can reduce CVD risk.

ELIGIBILITY:
Inclusion Criteria:

* Receiving primary care from participating physicians from practices in the Duke Primary Care Research Consortium
* Hypertension

Exclusion Criteria:

* Primary care doctor advises against enrollment
* Pregnant, nursing, or planning pregnancy
* Recent CVD event
* Chronic kidney or liver disease
* Active cancer

Min Age: 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 574 (Actual)
Dates: Start 2004-02; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

PRIMARY OUTCOMES:
Change in systolic blood pressure | 6 months

SECONDARY OUTCOMES:
Change in diastolic BP | 6 months
Change in BP at 18 months | 18 months
Patient and MD adherence to intervention | 6 and 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Laura P. Svetkey, Study Chair — Duke University
Locations (1):
- Duke University, Durham, North Carolina, United States

REFERENCES:
- [Derived] Svetkey LP, Pollak KI, Yancy WS Jr, Dolor RJ, Batch BC, Samsa G, Matchar DB, Lin PH. Hypertension improvement project: randomized trial of quality improvement for physicians and lifestyle modification for patients. Hypertension. 2009 Dec;54(6):1226-33. doi: 10.1161/HYPERTENSIONAHA.109.134874. PMID 19920081
- [Derived] Dolor RJ, Yancy WS Jr, Owen WF, Matchar DB, Samsa GP, Pollak KI, Lin PH, Ard JD, Prempeh M, McGuire HL, Batch BC, Fan W, Svetkey LP. Hypertension Improvement Project (HIP): study protocol and implementation challenges. Trials. 2009 Feb 26;10:13. doi: 10.1186/1745-6215-10-13. PMID 19245692